CLINICAL TRIAL: NCT05611190
Title: Coronary CT Angiography-Derived Fractional Flow Reserve-guided Optimize Treatment Strategy for In-stent Restenosis
Brief Title: CT-FFR-guided Strategy for In-stent Restenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yan'an Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: In-stent Restenosis
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease; In-stent Restenosis
Keywords: Coronary CT Angiography-derived Fractional Flow Reserve; In-stent Restenosis; Major Adverse Coronary Events
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Other): Participants randomized to usual care will be evaluated according to institutional standard practice. The investigators will review clinical data and results of the diagnostic tests to recommend a treatment strategy, according to the institution's standard practice.
  Interventions: Diagnostic Test: Usual Care
- CT-FFR (Experimental): Participants randomized to a CT-FFR strategy will be assigned to non-invasive CT-FFR evaluation. The investigators will review the results CT-FFR, and will recommend a further ICA test if CT-FFR≤0.8. The investigators will review the results of all available diagnostic tests, including CT-FFR and ICA, and will recommend a treatment strategy accordingly.
  Interventions: Diagnostic Test: CT-FFR

INTERVENTIONS:
Diagnostic Test: CT-FFR — CT-FFR is a type of non-invasive procedure to provide a 3D model of coronary arteries as a way to evaluate the hemodynamic significance of coronary artery lesions. CT-FFR calculates FFR from subject-specific CCTA data using computational fluid dynamics technology. CT-FFR value ≤0.80 is considered hemodynamically significant.
  Arms: CT-FFR
Diagnostic Test: Usual Care — Participants randomized to usual care will be evaluated according to institutional standard practice.
  Arms: Usual Care

SUMMARY:
This study will be a prospective, randomized clinical trial to compare standard practice guided by usual care testing to CT-FFR-guided management in patients with in-stent restenosis.

DETAILED DESCRIPTION:
This trial will randomize 294 patients with in-stent restenosis to receive either CT-FFR or routine clinical assessment. In all subjects, the investigators will review all diagnostic test results and determine a treatment strategy. The primary end point will be 12-month Major Adverse Coronary Event (MACE) rates, defined as all cause death, non-fatal myocardial infarction (MI), ischemia-driven target vessel revascularization (TVR). Secondary end points will include total medical costs, and quality of life (QOL), medical radiation exposure, etc. We will test noninferiority of current FFR-guided strategy compared with standard care strategy.

ELIGIBILITY:
Inclusion Criteria:

* (1) >18 years old;
* (2) ability to provide informed consent;
* (3) previous PCI who underwent CCTA and have at least 1 lesion with a percent diameter in-stent stenosis between 30% and 90% in a coronary artery with a ≥2.25 mm reference vessel diameter by visual assessment;
* (4) accepted further clinically indicated coronary testing, coronary arteriography, or FFR, or IVUS, or PCI, etc.

Exclusion Criteria:

* (1) Prior coronary artery bypass surgery (CABG), heart valve surgery, cardiac pacemaker, or implanted cardiac defibrillator;
* (2) Target vascular stents were evaluated for implantation within one month;
* (3) unstable clinical conditions including acute chest pain, cardiogenic shock, congestive heart failure (NYHA grade III or IV), unstable blood pressure (systolic blood pressure < 90mmHg) or acute pulmonary edema;
* (4) Acute myocardial infarction occurred within 7 days before enrollment, and left ventricular ejection fraction ≤40%;
* (5) Other severe cases are not suitable for clinical trials including complex congenital heart disease, sick sinus syndrome, long QT syndrome, severe arrhythmia, tachycardia, severe asthma, severe or very severe chronic obstructive pulmonary disease (COPD) and severe chronic renal damage;
* (6) Contraindication to beta blockers, nitroglycerin, adenosine, or allergy to iodine contrast agents;
* (7) Pregnancy or pregnancy status unknown;
* (8) Life expectancy <1 years;
* (9)Repeated enrollment;
* (10) Any other factors that other researchers consider not suitable for inclusion or completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2022-12-12 (Estimated); Primary Completion 2024-12-11 (Estimated); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
12-month MACE | 12 months
  12-month Major Adverse Coronary Event (MACE) rates, defined as:
  1. All cause death
  2. Non-fatal myocardial infarction (MI)
  3. Ischemia-driven target vessel revascularization (TVR)

SECONDARY OUTCOMES:
MACE | 3-month, 6-month, 24-month, 36-month
  MACE defined as:
  1. All cause death
  2. Non-fatal MI
  3. Clinical-driven TVR
Rates of Target lesion failure (TLF) | 3-month, 6-month, 24-month, 36-month
  Composite of clinically driven TLR, MI or cardiac death related to the target vessel.
Total costs | 6-month, 12-month
  Total costs will be calculated from the use of all cardiac-related invasive and non-invasive tests, revascularization procedures, hospital admissions and outpatient attendances due to a cardiovascular cause, and cardiac medications.
Quality of life (QOL) will be assessed using the EQ-5D-VAS questionnaire | 6-month, 12-month
  Quality of life (QOL), will be assessed using the EQ-5D-VAS questionnaire
Seattle Angina Questionnaire | 6-month, 12-month
  angina status, will be assessed using the Seattle Angina Questionnaire
Cumulative radiation exposure | 6-month, 12-month
  Cumulative radiation exposure within 6-month and 12-month of study entry included all cardiovascular tests and invasive procedures, including CTA, myocardial perfusion imaging, and ICA.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xue, Principal Investigator — Yan'an Affiliated Hospital of Kunming Medical University

IPD SHARING:
Plan to Share IPD: No